CLINICAL TRIAL: NCT02429505
Title: Treatment of Leishmaniasis With Impavido® (Miltefosine): Higher-Weight Patient Registry
Status: Withdrawn | Type: Observational
Why Stopped: This study was COMPLETED, but no patients were enrolled.
Sponsor: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: IMP 2127-4
Record Dates: First submitted 2015-04-22; First posted 2015-04-29 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Miltefosine: Miltefosine : target of 2.5 mg/kg/day for 28 days. Patients 45 kg or greater were to receive one 50 mg capsule 3 times daily for 28 consecutive days. This prospective observational study in which patients undergoing treatment for leishmaniasis with miltefosine in the United States who weighed >75 kg could volunteer to provide information about their clinical response to treatment up to 6 months after the start of treatment.
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — miltefosine: target 2.5 mg/kg/day for 28 days
  Other Names: Impavido

SUMMARY:
This study is a prospective observational study in which patients undergoing treatment for leishmaniasis with miltefosine (Impavido) in the US and who weigh > 75 kg can volunteer to provide information about their clinical response to treatment up to 6 months after the start of treatment.

DETAILED DESCRIPTION:
Objective: The purpose of this observational study is to fulfill PMR 2127-4 for the miltefosine NDA (204684): implement a higher-weight-patient registry for the time period Mar 2015-Mar 2020.

Study Design: This study is a prospective observational study in which patients undergoing treatment for leishmaniasis with Impavido in the US and who weigh > 75 kg can volunteer to provide information about their clinical response to treatment up to 6 months after the start of treatment.

Population: Leishmaniasis patients treated with Impavido who weigh more than 75 kg.

Drug Product:

Drug name: Impavido (50 mg capsules). Dosing regimen: as per the Impavido Product Label

Study Procedures: Patients who weigh more than 75 kg will become aware of the Impavido Higher-Weight Patient Registry via the Impavido website. By calling 1-866-588-5405, the patient will be connected to the Impavido Higher-Weight Patient Registry Coordinating Center. A trained staff member will acquaint the patient with the goals and procedures of the study. If the patient tentatively agrees to participate in the study over the telephone, the patient will be mailed information forms, the Consent/Assent Forms, and the Consent for the patient's physician to release medical information. Receipt of the two signed Consent and/or Assent Forms by the Coordinating Center will signify patient consent. The Coordinating Center will contact the patient's physician at the end of treatment, and at 1, 3, and 6 months after completing treatment, to collect data on efficacy and adverse effects (only during treatment).

Sample Size and Study Duration: Estimated 3-10 patients per year for 5 years.

Outcome Parameters:

Efficacy Adverse effects

Analysis: Baseline data, compliance to prescribed treatment, and outcomes will be reported for individual patients and for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Did the subject give consent to collect data from her or her physician?
2. Was the subject treated for leishmaniasis with miltefosine?
3. Does the subject weigh more than 75 kg?

Exclusion Criteria:

[none]

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: leishmaniasis patients who are administered miltefosine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Number of patients cured | 6 months
  Determination of possible relationship of lower mg/kg daily doses of miltefosine and efficacy

SECONDARY OUTCOMES:
Number of patients with adverse effects | 6 months
  Adverse events including symptoms and laboratory parameters (if available)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Ransom, PhD, Principal Investigator — Fast Track Drugs and Biologics LLC
Locations (1):
- Fast-Track Drugs and Biologics, LLC, Poolesville, Maryland, United States

DOCUMENTS (1):
  • Study Protocol (2014-12-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT02429505/Prot_000.pdf